CLINICAL TRIAL: NCT06560086
Title: Ketoconazole Contributes to Cryptorchidism Outcome Via Modulating Testicular Macrophage Trem2
Brief Title: Ketoconazole Contributes to Cryptorchidism Outcome Via Modulating Macrophage Trem2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 82171587
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-02

CONDITIONS: Cryptorchidism
Keywords: cryptorchidism; testicular macrophages; Leydig cells; immune micro-environment
MeSH Terms: conditions — Cryptorchidism | interventions — Ketoconazole; Luteinizing Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intact aborted fetal testicular tissue treated with ketoconazole (Experimental): A fetal developmental stage is precisely determined. Then, fetal tissues are extracted for in vitro cultivation. Intact aborted fetal testicular tissues are cultured in a medium containing 10-6 mol/L ketoconazole, which is the injectable solution powder. Ketoconazole is administered starting on the first day and then every other day, for a total of 7 times over the 14-day in vitro culture period.
  Interventions: Drug: Ketoconazole
- Intact aborted fetal testicular tissue treated with luteinizing hormone (Experimental): A fetal developmental stage is precisely determined. Then, fetal tissues are extracted for in vitro cultivation. Intact aborted fetal testicular tissues are cultured in a medium containing 1 IU/mL luteinizing hormone, which is the injectable solution powder. Luteinizing hormone is administered starting on the first day and then every other day, for a total of 7 times over the 14-day in vitro culture period.
  Interventions: Drug: Luteinizing Hormone
- Intact aborted fetal testicular tissue treated with none (No Intervention): A fetal developmental stage is precisely determined. Then, fetal tissues are extracted for in vitro cultivation. Intact aborted fetal testicular tissues are cultured in a medium.

INTERVENTIONS:
Drug: Ketoconazole — A fetal developmental stage is precisely determined. Then, fetal tissues are extracted for in vitro cultivation. Intact aborted fetal testicular tissues are cultured in a medium containing 10-6 mol/L ketoconazole, which is the injectable solution powder. Ketoconazole is administered starting on the first day and then every other day, for a total of 7 times over the 14-day in vitro culture period.
  Arms: Intact aborted fetal testicular tissue treated with ketoconazole
Drug: Luteinizing Hormone — A fetal developmental stage is precisely determined. Then, fetal tissues are extracted for in vitro cultivation. Intact aborted fetal testicular tissues are cultured in a medium containing 1 IU/mL luteinizing hormone, which is the injectable solution powder. Luteinizing hormone is administered starting on the first day and then every other day, for a total of 7 times over the 14-day in vitro culture period.
  Arms: Intact aborted fetal testicular tissue treated with luteinizing hormone

SUMMARY:
Reduced hormone insulin-like 3, exclusively secreted by Leydig cells, has been identified as the recognized mechanism for cryptorchidism. Testicular macrophages residing in the testicular interstitium were thought to play a vital role in maintaining hormone secretion of Leydig cells. However, the contribution of macrophages to cryptorchidism remained poorly understood. Here, after 14 days of ketoconazole treatment, levels of both Trem2 and insulin-like 3 significantly decrease in human embryonic testes compared to the untreated control group. Conversely, 14 days of luteinizing hormone stimulation lead to elevated levels of Trem2 and insulin-like 3 in the testes compared to the untreated control group. Additionally, researchers find a positive correlation between Trem2 and insulin-like 3 expression in a human ex vivo tissue culture model. In summary, the study will propose Trem2 as a novel target for maintaining normal testicular descent by regulating the testicular immune microenvironment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Termination of pregnancy is not related to the health of the fetus.
* 2. The fetus is intact in development and free of malformations and abnormalities.
* 3. Estimation of gestational age based on parietal-rump length must be between 8 and 13 weeks of gestation.

Exclusion Criteria:

* 1. The termination of pregnancy is related to the health of the fetus
* 2. The fetus is not intact in development.
* 3. The fetus has malformations, abnormalities
* 4. Estimation of gestational age based on parietal-rump length must not be within 8-13 weeks of gestation.

Ages: 8 Weeks to 13 Weeks | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-02-03 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Relative expression of Trem2 and insulin-like 3 protein | The date of 14 days cultured
  Ketoconazole promotes a decrease in Trem2 and a decrease in insulin-like 3, and they are strongly correlated.

CONTACTS AND LOCATIONS:
Overall Officials: Wenliang Ge, Study Director — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated hospital of nantong university, Nantong, Jiangsu, China